CLINICAL TRIAL: NCT00280254
Title: A Hemodynamically Oriented Echocardiography-Based Strategy in the Treatment of Congestive Heart Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Hospital de Clinicas de Porto Alegre (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCPA-ICC01
Record Dates: First submitted 2006-01-19; First posted 2006-01-20 (Estimated); Last update posted 2006-01-20 (Estimated); Status verified 2006-01

CONDITIONS: Heart Failure
Keywords: Heart Failure; Hemodynamics; Echocardiography
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Procedure: Hemodynamically Oriented Echocardiography-based Strategy

SUMMARY:
The purpose of this study was to compare two strategies in the treatment of outpatients with heart failure. We hypothesized that an individualized treatment strategy based on the availability of hemodynamic data from non-invasive testing would be feasible and significantly reduce morbidity compared to the conventional clinically oriented treatment of heart failure outpatients.

DETAILED DESCRIPTION:
Clinical strategies aiming at achieving an optimal hemodynamic profile have been advocated for the management of congestive heart failure. Non-invasive estimates, based on echocardiographic evaluations, might identify outpatients that could benefit from additional pharmacological therapy. Based on this assumption we conducted a single-center, prospective, randomized, open-label, blinded endpoint evaluation clinical trial comparing an echocardiography-guided strategy aimed at achieving a near-normal hemodynamic profile and the conventional clinically-oriented strategy for congestive heart failure management.

Echocardiography-guided strategy. Patients allocated to the echocardiography-guided strategy underwent sequential cardiac ultrasound examinations to evaluate hemodynamic-derived parameters. M-mode and two-dimensional color Doppler echocardiography was performed by an experienced cardiologist using commercially available ultrasound equipments (ATL HDI 5000, Bothel, WA, USA). Echocardiographic parameters were evaluated according to standard recommendations of the American Society of Echocardiography. For each measurement, 3-5 consecutive cardiac cycles were measured and averaged. Hemodynamic parameters were determined according to previously validated protocols. In brief, pulmonary artery systolic pressure was estimated as the sum of the estimated right atrial pressure and the pressure gradient between the right ventricle and right atria. Right atrial pressure was estimated by measuring the inferior vena cava diameter and its degree of collapsibility during inspiration. Cardiac output was determined by multiplying heart rate by left ventricular systolic volume. Left ventricular systolic volume was estimated by multiplying the time-velocity integral of the left ventricular outflow by the estimated left ventricular outflow area. Systemic vascular resistance was calculated using standard hemodynamic formulas, incorporating cardiac output and mean arterial pressure estimations. Systemic vascular resistance and cardiac output were indexed by body surface area. Each patient assigned to the echocardiography-guided strategy underwent three consecutive echocardiograms separated by four-week periods and a final echocardiogram at 6 months. Following each test, all patients were reevaluated by physicians from the heart failure team. Pharmacological therapy was then guided according to a pre-defined protocol based on hemodynamic estimates. Firstly, whenever elevated right-sided filling pressures were detected loop diuretic therapy was incremented irrespective of the presence of clinical signs and symptoms of pulmonary and/or systemic congestion. Afterwards, whenever raised systemic vascular resistance was identified, additional vasodilator therapy was incorporated or optimized, as long as systolic arterial pressure was equal or greater than 90 mmHg.

Clinically-guided strategy. Therapeutic decisions for patients assigned to the conventional treatment were based on recommendations from international clinical practice guidelines. Angiotensin converting enzyme inhibitors and beta-blockers use and optimization were encouraged. Standard non-pharmacological counseling was also provided by CHF trained nurses during the first month of follow-up. Diuretic therapy was exclusively based on the presence and intensity of clinical findings suggestive of pulmonary and/or systemic congestion. Clinically oriented patients also underwent a baseline and a final echocardiogram, but the decision-making team was unaware of this data throughout the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. age greater than 18 years old,
2. CHF diagnosis for more than 6 months regardless of etiology,
3. echocardiography-based left ventricular ejection fraction equal or less than 40%, and
4. prior CHF admission within three months from randomization

Exclusion Criteria:

1. thoracic deformity or severe chronic lung disease imposing technical limitation to perform high-quality echocardiography,
2. acute coronary syndrome in the last three months,
3. congenital heart disease,
4. moderate to severe stenotic heart valve disease or
5. end-stage renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102
Dates: Start 1999-11; Study Completion 2004-12

PRIMARY OUTCOMES:
The primary efficacy end-point was time to the first event of combined all-cause mortality and all-cause hospitalization or emergency room visit

SECONDARY OUTCOMES:
Secondary end-points were changes in hemodynamic estimates (right atrial pressure, systolic pulmonary artery pressure and systemic vascular resistance), serum electrolytic measurement and renal function.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine O Clausell, MD, Principal Investigator — Federal University of Rio Grande do Sul. Medical School